CLINICAL TRIAL: NCT05592795
Title: Explore the Effects and Mechanisms of ERCP and EST on Biliary Microecology
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Qi-Yong Li (Other)
Responsible Party: Sponsor-Investigator, Qi-Yong Li, professor, Shulan (Hangzhou) Hospital
Organization: Shulan (Hangzhou) Hospital (Other)
Other Study IDs: shulan(hangzhou)1
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Cholangiopancreatography, Endoscopic Retrograde; Choledocholithiasis; Gallstones
MeSH Terms: conditions — Choledocholithiasis; Gallstones

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples With DNA — microorganisms in bile
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with Gallbladder polyp or gallbladder adenomyosis: Patients with Gallbladder polyp or gallbladder adenomyosis In view of the difficulty in obtaining bile from normal people, our research team plans to select bile samples from patients undergoing laparoscopic cholecystectomy and patients with pathological diagnosis of gallbladder polyps or gallbladder adenomyosis as physiological bile of normal people.
- Patients with choledocholithiasis: Patients with choledocholithiasis The research group plans to select bile samples from patients with first episode choledocholithiasis, patients receiving ERCP treatment for the first time, and patients undergoing duodenal papillary incision during EST operation to study the biliary flora of patients with choledocholithiasis. Compared with the normal group, analyze whether there are differences, similarities and uniqueness between the groups, dynamically track changes in the structure of biliary flora before and after treatment, and whether there is specific flora related to the type of disease, and compared with the existing biliary microbiome database, to study whether there are new bacterial species.
  Interventions: Other: Whether ERCP or EST is carried out
- Patients with previous ERCP and/or EST operations and duodenal papilla incision during operation: Patients with previous ERCP and/or EST operations and duodenal papilla incision during operation Bile from patients who had undergone ERCP and EST duodenal papillary incision was collected, and the long-term impact of duodenal papillary incision on biliary microecology was discussed by comparing with that of normal patients.
  Interventions: Other: Whether ERCP or EST is carried out

INTERVENTIONS:
Other: Whether ERCP or EST is carried out — This project systematically studies the physiological characteristics of biliary microecology in normal people, and explores the impact of ERCP and EST duodenal papillary incision on biliary microecology.
  Groups: Patients with choledocholithiasis; Patients with previous ERCP and/or EST operations and duodenal papilla incision during operation

SUMMARY:
The objective of this observational study is to explore the structure of biliary flora in normal people, explore the dynamic impact of ERCP and EST on biliary microecology, study the marker flora, metabolites and functional genes related to biliary diseases, explore the occurrence and development mechanism, regulatory pathways and key targets of biliary diseases, and provide new strategies for the prevention and treatment of biliary diseases from the perspective of biliary microecology.

DETAILED DESCRIPTION:
Our research group applied the technology of macro genome sequencing to explore the biliary microecology through genomics and metabonomics analysis, describe the biliary microecology map of normal people, and build the biliary microecology framework of normal people; To explore the dynamic impact of ERCP and EST treatment on biliary tract microecology, and to further study the dynamic changes, abundance information and diversity characteristics of biliary tract microecology in patients with duodenal papillary incision and Oddi sphincter dysfunction, so as to find the marker flora and metabolites related to bile duct diseases, as well as the prognostic predictive value of specific flora and clinical diagnosis and treatment plan. This study provides a new direction for exploring the composition of human biliary microecology and the occurrence and development mechanism of biliary diseases and provides a new strategy for the treatment of patients with biliary diseases. It has important scientific significance and clinical value.

This project systematically studies the physiological characteristics of biliary tract microecology in normal people, explores the impact of ERCP and EST duodenal papillary incision on biliary tract microecology, clarifies the integrated genomic and metabolomic maps of biliary tract microorganisms in different states, compares the differences of biliary tract microecology at different key nodes, looks for the marker flora related to ERCP and EST treatment, and analyzes the correlation between the marker flora and clinical characteristics, To explore the role and mechanism of key bacteria in the occurrence and development of biliary diseases, so as to provide theoretical basis and strategies for improving prognosis for clinical treatment.

Purpose of this study

1. To construct the framework of biliary microecology in normal people, and define the structure and metabolite characteristics of biliary flora;
2. To study the short-term and long-term changes of biliary microecology in patients with ERCP, EST duodenal papillary incision and Oddi sphincter dysfunction, and explore the influence of specific pathogenic bacteria on the occurrence and development of biliary diseases
3. To screen the key flora of biliary microecology disorder before and after ERCP and EST treatment, and to explore the role and mechanism of marker flora in the occurrence and development of biliary diseases.

ELIGIBILITY:
1.Patients with Gallbladder polyp or gallbladder adenomyosis:

Inclusion Criteria:

1. The patient received laparoscopic cholecystectomy in our hospital from September 1, 2022 to September 1, 2023;
2. Age>18 years old;
3. Postoperative pathology was gallbladder polyp or gallbladder adenomyosis.

Exclusion Criteria:

1. Preoperative biliary surgery history or intraoperative biliary injuried;
2. Other complications were found.

2.Patients with choledocholithiasis:

Inclusion Criteria:

1. The patients were treated in our center from September 1, 2022 to September 1, 2023;
2. Age>18 years old;
3. Patients with choledocholithiasis received ERCP and EST treatment for the first time, but did not receive treatment in other hospitals;
4. The nasobiliary duct is to be retained to drain bile.

Exclusion Criteria:

1. Acute cholangitis;
2. There are serious complications.

3.Patients with previous ERCP and/or EST operations and duodenal papilla incision during operation:

Inclusion Criteria:

1. The patients received ERCP treatment in our center from September 1, 2022 to September 1, 2023;
2. Age>18 years old;
3. He has had ERCP and EST operations in the past, and the duodenal papilla was cut during the operation;

Exclusion Criteria:

1. Acute cholangitis;
2. Serious complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients with Gallbladder polyp or gallbladder adenomyosis
  2. Patients with choledocholithiasis
  3. Patients with previous ERCP and/or EST operations and duodenal papilla incision during operation
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Successfully collect all bile samples required | 1 week
  Collect the required bile samples under the required conditions according to the difference of the three groups.Then DNA extraction, Illumina MiSeq sequencing and bioinformatics analysis will be performed on the collected samples.

CONTACTS AND LOCATIONS:
Overall Officials: Qi-Yong Li, doctor, Study Director — Shulan (Hangzhou) Hospital
Locations (3):
- China (3):
  - Shulan (Hangzhou) Hospital, Hangzhou, Zhejiang
  - Quzhou People's Hospital, Quzhou, Zhejiang
  - Shulan (Quzhou) Hospital, Quzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Konturek PC, Haziri D, Brzozowski T, Hess T, Heyman S, Kwiecien S, Konturek SJ, Koziel J. Emerging role of fecal microbiota therapy in the treatment of gastrointestinal and extra-gastrointestinal diseases. J Physiol Pharmacol. 2015 Aug;66(4):483-91. PMID 26348073
- [Background] Yu LX, Schwabe RF. The gut microbiome and liver cancer: mechanisms and clinical translation. Nat Rev Gastroenterol Hepatol. 2017 Sep;14(9):527-539. doi: 10.1038/nrgastro.2017.72. Epub 2017 Jul 5. PMID 28676707
- [Background] Mima K, Nakagawa S, Sawayama H, Ishimoto T, Imai K, Iwatsuki M, Hashimoto D, Baba Y, Yamashita YI, Yoshida N, Chikamoto A, Baba H. The microbiome and hepatobiliary-pancreatic cancers. Cancer Lett. 2017 Aug 28;402:9-15. doi: 10.1016/j.canlet.2017.05.001. Epub 2017 May 17. PMID 28527946
- [Background] Molinero N, Ruiz L, Milani C, Gutierrez-Diaz I, Sanchez B, Mangifesta M, Segura J, Cambero I, Campelo AB, Garcia-Bernardo CM, Cabrera A, Rodriguez JI, Gonzalez S, Rodriguez JM, Ventura M, Delgado S, Margolles A. The human gallbladder microbiome is related to the physiological state and the biliary metabolic profile. Microbiome. 2019 Jul 4;7(1):100. doi: 10.1186/s40168-019-0712-8. PMID 31272480
- [Background] Shen H, Ye F, Xie L, Yang J, Li Z, Xu P, Meng F, Li L, Chen Y, Bo X, Ni M, Zhang X. Metagenomic sequencing of bile from gallstone patients to identify different microbial community patterns and novel biliary bacteria. Sci Rep. 2015 Dec 2;5:17450. doi: 10.1038/srep17450. PMID 26625708
- [Background] Ye F, Shen H, Li Z, Meng F, Li L, Yang J, Chen Y, Bo X, Zhang X, Ni M. Influence of the Biliary System on Biliary Bacteria Revealed by Bacterial Communities of the Human Biliary and Upper Digestive Tracts. PLoS One. 2016 Mar 1;11(3):e0150519. doi: 10.1371/journal.pone.0150519. eCollection 2016. PMID 26930491
- [Background] Swidsinski A, Ludwig W, Pahlig H, Priem F. Molecular genetic evidence of bacterial colonization of cholesterol gallstones. Gastroenterology. 1995 Mar;108(3):860-4. doi: 10.1016/0016-5085(95)90461-1. PMID 7875489
- [Background] Kawai M, Iwahashi M, Uchiyama K, Ochiai M, Tanimura H, Yamaue H. Gram-positive cocci are associated with the formation of completely pure cholesterol stones. Am J Gastroenterol. 2002 Jan;97(1):83-8. doi: 10.1111/j.1572-0241.2002.05425.x. PMID 11808974
- [Background] Kose SH, Grice K, Orsi WD, Ballal M, Coolen MJL. Metagenomics of pigmented and cholesterol gallstones: the putative role of bacteria. Sci Rep. 2018 Jul 25;8(1):11218. doi: 10.1038/s41598-018-29571-8. PMID 30046045
- [Background] Law R, Baron TH. ERCP. Gastrointest Endosc. 2013 Sep;78(3):428-33. doi: 10.1016/j.gie.2013.06.018. No abstract available. PMID 23948191
- [Background] Li QY, Pan L, Ling Q, He JD, Zhang LX, Zheng SS. Single-operator wire-guided cannulation technique enables easier cannulation of endoscopic retrograde cholangiopancreatography. Dig Dis Sci. 2012 Dec;57(12):3293-8. doi: 10.1007/s10620-012-2274-5. Epub 2012 Jun 27. PMID 22736016
- [Background] Li QY, Chen KJ, Jin J, Zheng SS. Guide wire-assisted technique to access the bile duct with biopsy forceps for repositioning and removal of metal stents. Endoscopy. 2013;45 Suppl 2 UCTN:E273-4. doi: 10.1055/s-0033-1344591. Epub 2013 Sep 5. No abstract available. PMID 24008462
- [Background] Williams EJ, Green J, Beckingham I, Parks R, Martin D, Lombard M; British Society of Gastroenterology. Guidelines on the management of common bile duct stones (CBDS). Gut. 2008 Jul;57(7):1004-21. doi: 10.1136/gut.2007.121657. Epub 2008 Mar 5. PMID 18321943
- [Background] Saito H, Kadono Y, Shono T, Kamikawa K, Urata A, Nasu J, Imamura H, Matsushita I, Tada S. Remaining issues of recommended management in current guidelines for asymptomatic common bile duct stones. World J Gastroenterol. 2021 May 14;27(18):2131-2140. doi: 10.3748/wjg.v27.i18.2131. PMID 34025069
- [Background] Kageoka M, Watanabe F, Maruyama Y, Nagata K, Ohata A, Noda Y, Miwa I, Ikeya K. Long-term prognosis of patients after endoscopic sphincterotomy for choledocholithiasis. Dig Endosc. 2009 Jul;21(3):170-5. doi: 10.1111/j.1443-1661.2009.00880.x. PMID 19691764